## Yellow Micropulse Laser 577-nm vs Infrared Diode Micropulse Laser 810-nm For the Treatment of Diabetic Macular Edema

Statistical analysis plan

12-10-2017

## Statistical Analysis:

Data were collected, revised, coded and entered to the Statistical Package for Social Science (IBM SPSS) version 23. The quantitative data were presented as mean, standard deviations and ranges when their distribution found parametric and median with inter-quartile range (IQR) when their distribution found non parametric. Qualitative variables were presented as number and percentages. The comparison between groups regarding qualitative data was done by using Chi-square test. The comparison between two paired groups with quantitative data and parametric distribution were done by using Paired ttest. While comparison between more than two paired groups with quantitative data and parametric distribution were done by using repeated measure ANOVA test. The comparison between two paired groups with quantitative data and non-parametric distribution were done by using Wilcoxon Rank test. While comparison between more than two paired groups with quantitative data and non-parametric distribution were done by using Friedman test. The confidence interval was set to 95% and the margin of error accepted was set to 5%. So, the p-value was considered significant as the following: P-value > 0.05: Non significant (NS), P-value < 0.05: Significant (S) and P-value < 0.01: Highly significant (HS).